CLINICAL TRIAL: NCT00329407
Title: The Effects of Topiramate on Alcohol Use in Alcohol Dependent Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Ofra Sarid-Segal, MD, Boston University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-22296
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Results first posted 2010-08-04 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-08

CONDITIONS: Alcoholism
Keywords: Alcoholism; Heavy Drinking; Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Topiramate

ARMS (1):
- Topiramate Treatment (Active Comparator): In this open label non-placebo controlled trial all subjects received topiramate, the active medication. Medication Dosing Schedule: Days 1-3 50 mg q PM Days 4-7 50 mg BID Days 8-11 50 mg q AM & 100 mg q PM Days 12-15 100mg BID Days 16-19 100 mg q AM & 150 mg q PM Days 20-23 150 mg BID Days 24-27 150 mg qAM & 200 mg q PM Days 28-70 200 mg BID Days 71-77 150 mg BID Days 78-84 100mg BID Days 85-87 50 mg BID Days 88-91 50 mg qPM
  Interventions: Drug: Topiramate (Topamax)

INTERVENTIONS:
Drug: Topiramate (Topamax) — Medication Dosing Schedule: Days 1-3 50 mg q PM Days 4-7 50 mg BID Days 8-11 50 mg q AM & 100 mg q PM Days 12-15 100mg BID Days 16-19 100 mg q AM & 150 mg q PM Days 20-23 150 mg BID Days 24-27 150 mg qAM & 200 mg q PM Days 28-70 200 mg BID Days 71-77 150 mg BID Days 78-84 100mg BID Days 85-87 50 mg BID Days 88-91 50 mg qPM

SUMMARY:
This investigation will assess the effectiveness of topiramate in reducing ethanol consumption by alcohol dependent subjects. It also will seek to establish whether topiramate can be safely used in this population including whether it might be subject to abuse by alcohol dependent individuals.

A secondary goal of this study is to assess the effects of topiramate on verbal fluency during treatment for alcohol dependence.

DETAILED DESCRIPTION:
Alcoholism is a disorder that produces extensive morbidity and mortality. Substantial progress has been made in the development of medications that can help to promote abstinence in alcohol dependent individuals. However, investigations of the most promising drugs, particularly naltrexone and acamprosate, suggest that these agents have at best moderate efficacy and there is a great need for additional medications for the treatment of alcoholism.

The results of a recent study suggest that the administration of the anticonvulsant agent ,topiramate helps alcoholic individuals to maintain abstinence (Johnson et al., 2003). The objectives of this study is to determine whether topiramate will reduce the consumption of alcohol in subjects dependent on this substance, as has been previously reported.Other study objectives are to assess the abuse liability properties of topiramate in alcohol dependent subjects and to examine the effects of chronic topiramate administration on cognitive functioning.

This will be a thirteen week long open label clinical trial of the effects of topiramate administration on ethanol consumption by alcohol dependent subjects.

Subjects will be asked to provide informed consent and then will be screened on the same day to determine if they meet study eligibility criteria. Subjects will be asked to return to provide two urines over the following week.

Baseline measures of mood, craving, withdrawal, cognitive functioning and physical health will be obtained. In the afternoon they will receive their first dose of medication. Their responses to this medication challenge will be assessed over a 3-hour period.

During the drug treatment phase subjects will be asked to come to the clinic weekly for assessment and manual guided therapy during weeks 1-4 and biweekly during weeks 6-8. On day 85 subjects will be seen at the clinic for a termination visit.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV Diagnosis of Alcohol Dependence; Minimal drinking level of 14 drinks per week for women and 20 drinks per week for men over a consecutive 30 day period during the last 90 days
2. Intent to stop drinking
3. Male or female age 18-65
4. Able to maintain sobriety for 3 consecutive days without the use of detoxification medications
5. Able to provide informed consent and to comprehend study procedures.
6. If a woman, then is willing to use an effective means of birth control during throughout the study period. These include: a. barrier (diaphragm or condom) with spermicide b.intrauterine progesterone contraceptive system c. levonorgestrel implant d. medroxyprogesterone acetate contraceptive injection e. complete abstinence

Exclusion Criteria:

1. Dependent on or extensive abuse of drugs or substances other than ethanol, nicotine, or caffeine as assessed by urine toxicology (2 out of 3 Dependent on or extensive abuse of drugs or substances other than positive consecutive urines)
2. DSM IV Axis I diagnoses other than ethanol, caffeine, or nicotine dependence severe enough to require treatment with medication or to prevent compliance with the protocol.
3. Currently being treated with disulfiram (Antabuse), naltrexone (ReVia), or acamprosate
4. Currently being treated with any other psychoactive or other CNS medications or a carbonic anhydrase inhibitor (e.g. acetazolamide)
5. In need of medical detoxification from alcohol.
6. Prior history of kidney stones.
7. History of liver disease. ALT or AST 3 times higher than upper range of normal values.
8. BUN or serum creatinine outside the normal range
9. Major neurological disorder including seizures
10. Other major diseases including severe hypertension, renal disease, or cardiac disease.
11. Prior participation within 60 days in another clinical study.
12. If female, a positive serum HCG or breast feeding.
13. If female using oral contraceptives as a means of birth control.
14. History of allergic sensitivity to topiramate
15. Pending imprisonment
16. Cardiac pacemaker or metal surgical implant.
17. History of angle closure glaucoma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ofra Sarid-Segal, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Dept of Psychiatry Clinical Studies Unit, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate Treatment: In this open label non-placebo controlled trial all subjects received topiramate, the active medication.
Period: Overall Study
Arm/Group | Topiramate Treatment
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Topiramate Treatment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 50.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Will be Subjects Ethanol Consumption Over the Course of the Drug Treatment Period as Assessed by the Timeline Followback Method
Description: The primary outcome was the mean daily consumption of standard alcoholic drinks (14 g per ethanol) during the baseline week compared to week 10, the final week subjects were one maintenance dose of topirmate.
Time Frame: 70 days
Population: An ITT approach was used in the analysis. Least squares value for the baseline and 10 week of treatment were compared using a t test with Dunnett-Hsu adjustment. Differences between these means are presented as the result.
Measure: Mean (Standard Error); unit: Standard Drink (14 g alcohol)
Arm/Group | Topiramate Treatment
Number analyzed (Participants) | 10
Standard Drink (14 g alcohol) | -4.9 (0.86)
Statistical Analysis 1: Comparison: Topiramate Treatment; This was a within subject analysis. The null hypothesis was that there would be no significant difference in least squares means values obtained for the baseline and week 10 assessment weeks; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The Dunnett-Hsu adjustment was used to correct for multiple comparisons; Mean Difference (Final Values) = -4.7, 95% CI 2-sided [-6.58 to -3.14], Standard Error of Mean 0.8

2. Secondary Outcome: Phonetic Portion of the Controlled Word Association Test (COWAT)
Description: Phonetic COWAT is a measure of verbal fluency. Results are in terms of number of words produced starting with a set of particular letters.This involves a comparison of baseline and Week 10 COWAT scores
Time Frame: Baseline compared to Week 10
Measure: Mean (Standard Error); unit: Number of words
Arm/Group | Topiramate Treatment
Number analyzed (Participants) | 10
Number of words | -11 (2.7)
Statistical Analysis 1: Comparison: Topiramate Treatment; This is a within subject comparison of COWAT scores botained for the baseline session and the Week 10 session. The null hypothesis is that there would be no difference between these scores; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — There would a significant reduction in COWAT scores between baseline and Week 10; The Dunnett-Hsu adjustment was used to correct for multiple comparisons; Mean Difference (Net) = -11, Standard Error of Mean 2.7

ADVERSE EVENTS:
Arm/Group | Topiramate Treatment
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate Treatment (N=10)
Agitation and Impaired Concentration (Nervous system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Limitation of this trial include the small number of subjects included and lack of blinding, and inculsion of a placebo control group. An other limitation was the testing the active medication topiramate at om=nly one dose level (i.e. 400 mg daily).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes